CLINICAL TRIAL: NCT02230566
Title: A Randomized, Placebo-Controlled, Blind-Start, Single-Crossover Phase 3 Study to Assess the Efficacy and Safety of UX003 rhGUS Enzyme Replacement Therapy in Patients With MPS 7
Brief Title: A Phase 3 Study of UX003 Recombinant Human Betaglucuronidase (rhGUS) Enzyme Replacement Therapy in Patients With Mucopolysaccharidosis Type 7 (MPS 7)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UX003-CL301
Expanded Access: NCT03775174 (Available)
Record Dates: First submitted 2014-08-22; First posted 2014-09-03 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: MPS 7; Sly Syndrome; Mucopolysaccharidosis; MPS VII
Keywords: MPS 7; Sly Syndrome; Mucopolysaccharidosis; MPS VII; Enzyme Replacement Therapy; Mucopolysaccharidosis type 7; rare disease; lysosomal storage disease; metabolic disorder
MeSH Terms: conditions — Mucopolysaccharidosis VII; Mucopolysaccharidoses; Rare Diseases; Lysosomal Storage Diseases; Metabolic Diseases | interventions — vestronidase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A: 4 mg/kg UX003 (Experimental): 4 mg/kg UX003 QOW through Week 46
  Interventions: Drug: UX003
- Group B: 8 Weeks Placebo then 4 mg/kg UX003 (Experimental): Placebo QOW for the first 8 weeks followed by 4 mg/kg UX003 QOW through Week 46
  Interventions: Drug: UX003; Other: Placebo
- Group C: 16 Weeks Placebo then 4 mg/kg UX003 (Experimental): Placebo QOW for the first 16 weeks followed by 4 mg/kg UX003 QOW through Week 46
  Interventions: Drug: UX003; Other: Placebo
- Group D: 24 Weeks Placebo then 4 mg/kg UX003 (Experimental): Placebo QOW for the first 24 weeks followed by 4 mg/kg UX003 QOW through Week 46
  Interventions: Drug: UX003; Other: Placebo

INTERVENTIONS:
Drug: UX003 — UX003 is a sterile concentrate formulation of rhGUS for intravenous infusion
  Other Names: recombinant human beta-glucuronidase; rh-β-glucuronidase; rhGUS
Other: Placebo — Placebo consisting of the UX003 formulation buffer (without rhGUS)
  Other Names: Reference therapy
  Arms: Group B: 8 Weeks Placebo then 4 mg/kg UX003; Group C: 16 Weeks Placebo then 4 mg/kg UX003; Group D: 24 Weeks Placebo then 4 mg/kg UX003

SUMMARY:
The Phase 3 study will use a novel randomized, intra-subject placebo-controlled, single crossover design, referred to as Blind Start, to evaluate the safety and efficacy of UX003. The Blind Start is a novel design whereby participants will be randomized to 1 of 4 groups, each representing a different treatment sequence, and will cross over to UX003 at different pre-defined time points in a blinded manner. All groups will receive a minimum of 24 weeks treatment with 4 mg/kg UX003 every other week (QOW).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MPS 7 based on leukocyte or fibroblast glucuronidase enzyme assay or genetic testing.
* Elevated urinary glycosaminoglycan (uGAG) excretion at a minimum of 3-fold over the mean normal for age (at Screening).
* Apparent clinical signs of lysosomal storage disease as judged by the Investigator, including at least one of the following: enlarged liver and spleen, joint limitations, airway obstruction or pulmonary problems, limitation of mobility while still ambulatory.
* Aged 5 - 35 years, inclusive.
* Willing and able to provide written informed consent, or in the case of subjects under the age of 18 (or 16 years, depending on the region), provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures.
* Sexually active subjects must be willing to use acceptable highly effective methods of contraception while participating in the study and for 30 days following the last dose.
* Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have not experienced menarche, or have had tubal ligation at least one year prior to Screening, or who have had total hysterectomy.
* Naïve to treatment with UX003.

Exclusion Criteria:

* Undergone a successful bone marrow or stem cell transplant or has any degree of detectable chimaerism with donor cells.
* Major surgery within 3 months prior to study entry or planned major surgery during the study that may not allow safe participation in the study.
* Presence or history of any hypersensitivity to rhGUS or its excipients that, in the judgment of the Investigator, places the subject at increased risk for adverse effects.
* Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study.
* Use of any investigational product (drug or device or combination) within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Presence of a condition of such severity and acuity that, in the opinion of the Investigator, warrants immediate surgical intervention or other treatment or may not allow safe participation in the study.
* Concurrent disease or condition, or laboratory abnormality that, in the view of the Investigator, places the subject at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or introduce additional safety concerns.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Harmatz, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland; Raymond Wang, MD, Principal Investigator — Children's Hospital of Orange County; Mislen Bauer, MD, Principal Investigator — Nicklaus Children's Hospital f/k/a Miami Children's Hospital; Chester Whitley, MD, Principal Investigator — University of Minnesota
Locations (4):
- United States (4):
  - Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Miami Children's Hospital, Miami, Florida
  - University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- [Result] Wang RY, da Silva Franco JF, Lopez-Valdez J, Martins E, Sutton VR, Whitley CB, Zhang L, Cimms T, Marsden D, Jurecka A, Harmatz P. The long-term safety and efficacy of vestronidase alfa, rhGUS enzyme replacement therapy, in subjects with mucopolysaccharidosis VII. Mol Genet Metab. 2020 Mar;129(3):219-227. doi: 10.1016/j.ymgme.2020.01.003. Epub 2020 Jan 11. PMID 32063397
- [Result] Harmatz P, Whitley CB, Wang RY, Bauer M, Song W, Haller C, Kakkis E. A novel Blind Start study design to investigate vestronidase alfa for mucopolysaccharidosis VII, an ultra-rare genetic disease. Mol Genet Metab. 2018 Apr;123(4):488-494. doi: 10.1016/j.ymgme.2018.02.006. Epub 2018 Feb 12. PMID 29478819
- [Derived] Montano AM, Rozdzynska-Swiatkowska A, Jurecka A, Ramirez AN, Zhang L, Marsden D, Wang RY, Harmatz P. Growth patterns in patients with mucopolysaccharidosis VII. Mol Genet Metab Rep. 2023 Jun 26;36:100987. doi: 10.1016/j.ymgmr.2023.100987. eCollection 2023 Sep. PMID 37415957
- [Derived] Tandon PK, Kakkis ED. The multi-domain responder index: a novel analysis tool to capture a broader assessment of clinical benefit in heterogeneous complex rare diseases. Orphanet J Rare Dis. 2021 Apr 19;16(1):183. doi: 10.1186/s13023-021-01805-5. PMID 33874971
- [Derived] Qi Y, McKeever K, Taylor J, Haller C, Song W, Jones SA, Shi J. Pharmacokinetic and Pharmacodynamic Modeling to Optimize the Dose of Vestronidase Alfa, an Enzyme Replacement Therapy for Treatment of Patients with Mucopolysaccharidosis Type VII: Results from Three Trials. Clin Pharmacokinet. 2019 May;58(5):673-683. doi: 10.1007/s40262-018-0721-y. PMID 30467742

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: 4 mg/kg UX003: 4 mg/kg UX003 every other week (QOW) through Week 46
Period: Overall Study
Arm/Group | Group A: 4 mg/kg UX003 | Group B: 8 Weeks Placebo Then 4 mg/kg UX003 | Group C: 16 Weeks Placebo Then 4 mg/kg UX003 | Group D: 24 Weeks Placebo Then 4 mg/kg UX003
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: 4 mg/kg UX003 | Group B: 8 Weeks Placebo Then 4 mg/kg UX003 | Group C: 16 Weeks Placebo Then 4 mg/kg UX003 | Group D: 24 Weeks Placebo Then 4 mg/kg UX003 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.13 (1.656) | 12.50 (4.004) | 20.77 (3.004) | 15.23 (8.633) | 15.41 (5.492)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 0 | 8
  Male | 0 | 1 | 0 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: European Union (EU) and Rest of World: Percentage Change From Baseline in Urinary Glycosaminoglycan (uGAG) Dermatan Sulfate (DS) at UX003 Treatment Week 24
Description: Baseline was defined as the average of all assessments prior to or on the date of cross-over to active treatment with UX003. (This provides the valid assessment, as placebo effect was subtracted from the treatment effect estimate providing a more conservative assessment of the true treatment effect.) Percent change from baseline in uGAG DS was analyzed by generalized estimating equation (GEE) modeling based on observed data. The GEE model included included baseline value, and the UX003 treatment week as a categorical variable. The covariance structure within subjects was assumed to be exchangeable.
  In the United States (US), this was considered a secondary outcome measure. Per guidance from the Food and Drug Administration (FDA), no primary efficacy variable was declared in the US. Efficacy was to be based on the totality of the clinical data on a per participant basis.
Time Frame: Baseline (defined as the average of all assessments prior to or on the date of cross-over to active treatment with UX003) to 24 weeks of UX003 study drug treatment
Population: Participants who had non-missing baseline and ≥1 post-baseline value during 24 weeks of UX003 treatment. Given a randomized blind start and single crossover study design, all 4 groups received a minimum of 24 weeks of UX003 treatment, with a placebo treatment period ranging from 0-24 weeks, by group. Analysis of placebo data was not planned.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Groups:
- UX003 4 mg/kg: Participants were randomized 1:1:1:1 to 1 of 4 treatment sequence groups to either start treatment with 4 mg/kg UX003 (Group A), or placebo for the first 8 weeks (Group B), 16 weeks (Group C) or 24 weeks (Group D) of the study and cross over to 4 mg/kg UX003. Participants were dosed QOW through Week 46. All groups received a minimum of 24 weeks of treatment with 4 mg/kg UX003 QOW.
Arm/Group | UX003 4 mg/kg
Number analyzed (Participants) | 12
percentage change | -64.82 (2.468)
Statistical Analysis 1: Comparison: UX003 4 mg/kg; Test type: Superiority; p < 0.0001, GEE — P-values are from GEE model including baseline value, and the post UX003 Treatment Week as a categorical variable. The covariance structure within participants was assumed to be exchangeable; LS Mean = -64.82, 95% CI 2-sided [-69.66 to -59.98]

2. Secondary Outcome: Multi-Domain Responder Index (MDRI) Score at UX003 Treatment Week 24
Description: MDRI score, calculated as the total response score at UX003 Treatment Week 24 across 6 domains: 6-Minute Walk Test, forced vital capacity predicted value, shoulder flexion, visual acuity, and Bruininks-Oseretsky Test of Motor Proficiency fine motor and gross motor capacity. For each domain, a minimally important difference (MID) was pre-specified. Changes from before treatment (baseline) to 24 weeks after treatment in each domain variable were scored against pre-specified MIDs. (This provides the valid assessment, as placebo effect would be subtracted from the treatment effect estimate providing a more conservative assessment of the true treatment effect.) An improvement or decline ≥ MID was scored either as a +1 or -1, respectively, and a change <MID was scored as 0. The integration of benefit occurred by summing the responses (-1, +1, 0) across all 6 domain variables to derive the MDRI score, with a range of -6 (greatest possible decline) to +6 (greatest possible improvement).
Time Frame: Baseline (defined as the last assessment prior to or on the date of cross-over to active treatment with UX003) to 24 weeks of UX003 study drug treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UX003 4 mg/kg
Number analyzed (Participants) | 12
units on a scale | 0.5 (0.8)
Statistical Analysis 1: Comparison: UX003 4 mg/kg; Test type: Superiority; p = 0.0527, t-test; P value from t-test of "no change" (0 change) from baseline

3. Secondary Outcome: Change From Baseline in 6-Minute Walk Test (6MWT) at UX003 Treatment Week 24
Description: The total distance walked (in meters) in a 6-minute period was measured. Baseline was defined as the last assessment prior to or on the date of cross-over to active treatment with UX003. (This provides the valid assessment, as placebo effect would be subtracted from the treatment effect estimate providing a more conservative assessment of the true treatment effect.) A positive change from Baseline indicates improvement. Change from baseline in 6MWT was analyzed by GEE modeling based on observed data. The GEE model included all participants who had non-missing baseline and at least one post-baseline value during the 24 weeks of UX003 treatment. The model included baseline value, and the UX003 treatment week as a categorical variable. The covariance structure within participants was assumed to be exchangeable.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | UX003 4 mg/kg
Number analyzed (Participants) | 9
meters | 20.8 (16.75)
Statistical Analysis 1: Comparison: UX003 4 mg/kg; Test type: Superiority; p = 0.2137, GEE — [p-value comment as in outcome 1, analysis 1]; LS Mean = 20.8, 95% CI 2-sided [-12.0 to 53.7]

4. Secondary Outcome: Change From Baseline in Pulmonary Function Testing: Percentage of Predicted Forced Vital Capacity (FVC%Pred) at UX003 Treatment Week 24
Description: Spirometry was administered to participants who did not require invasive ventilatory support or have a tracheostomy and measured percentage of predicted FVC. The percent predicted values were calculated after testing using published normative data. Baseline was defined as the last assessment prior to or on the date of cross-over to active treatment with UX003. (This provides the valid assessment, as placebo effect would be subtracted from the treatment effect estimate providing a more conservative assessment of the true treatment effect.) No GEE analysis was performed for FVC due to the limitation of the sample size.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage predicted FVC
Arm/Group | UX003 4 mg/kg
Number analyzed (Participants) | 1
percentage predicted FVC | 0 (NA) — 1 participant evaluated

5. Secondary Outcome: Change From Baseline in Pulmonary Function Testing: Maximum Ventilatory Ventilation (MVV) at UX003 Treatment Week 24
Description: Spirometry was administered to participants who did not require invasive ventilatory support or have a tracheostomy to measure MVV. The percent predicted values were calculated after testing using published normative data. Baseline was defined as the last assessment prior to or on the date of cross-over to active treatment with UX003. (This provides the valid assessment, as placebo effect would be subtracted from the treatment effect estimate providing a more conservative assessment of the true treatment effect.)
Time Frame: as for outcome 2
Population: No change from baseline was calculated and no GEE analysis was performed due to lack of data at baseline and/or UX003 Treatment Week 24.
Arm/Group | UX003 4 mg/kg
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Shoulder Flexion and Extension Maximum Range of Motion at UX003 Treatment Week 24
Description: Goniometry was used to measure (in degrees) the maximum passive shoulder range of motion in both flexion and extension. Baseline was defined as the last assessment prior to or on the date of cross-over to active treatment with UX003. (This provides the valid assessment, as placebo effect would be subtracted from the treatment effect estimate providing a more conservative assessment of the true treatment effect.) Change from baseline in shoulder flexion-left was analyzed by GEE modeling based on observed data. The GEE model included all participants who had non-missing baseline and at least one post-baseline value during the 24 weeks of UX003 treatment. The model included baseline value, and the UX003 treatment week as a categorical variable. The covariance structure within participants was assumed to be exchangeable.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: degrees
Arm/Group | UX003 4 mg/kg
Number analyzed (Participants) | 12
degrees
  Shoulder flexion - left | -6.5 (4.86)
  Shoulder extension - left: number analyzed (Participants) | 11
  Shoulder extension - left | -1.5 (4.83)
  Shoulder flexion - right | -1.8 (3.54)
  Shoulder extension - right: number analyzed (Participants) | 11
  Shoulder extension - right | -3.4 (3.48)
  Tighter shoulder flexion | -9.4 (4.6)
  Tighter shoulder extension: number analyzed (Participants) | 11
  Tighter shoulder extension | -6.7 (3.53)
Statistical Analysis 1: Comparison: UX003 4 mg/kg; Shoulder Flexion - Left; Test type: Superiority; p = 0.1778, GEE; LS Mean = -6.5, 95% CI 2-sided [-16.1 to 3.0]
Statistical Analysis 2: Comparison: UX003 4 mg/kg; Shoulder Extension - Left; Test type: Superiority; p = 0.7632, GEE; LS Mean = -1.5, 95% CI 2-sided [-10.9 to 8.0]
Statistical Analysis 3: Comparison: UX003 4 mg/kg; Shoulder Flexion - Right; Test type: Superiority; p = 0.6034, GEE; LS Mean = -1.8, 95% CI 2-sided [-8.8 to 5.1]
Statistical Analysis 4: Comparison: UX003 4 mg/kg; Shoulder Extension - Right; Test type: Superiority; p = 0.3332, GEE; LS Mean = -3.4, 95% CI 2-sided [-10.2 to 3.4]
Statistical Analysis 5: Comparison: UX003 4 mg/kg; Tighter Shoulder Flexion; Test type: Superiority; p = 0.0415, GEE; LS Mean = -9.4, 95% CI 2-sided [-18.4 to -0.4]
Statistical Analysis 6: Comparison: UX003 4 mg/kg; Tighter Shoulder Extension; Test type: Superiority; p = 0.0563, GEE; LS Mean = -6.7, 95% CI 2-sided [-13.6 to 0.2]

7. Secondary Outcome: Change From Baseline in Uncorrected Visual Acuity at UX003 Treatment Week 24
Description: Visual acuity was measured (corrected and uncorrected) using a standard eye chart and recorded for each eye independently. Baseline was defined as the last assessment prior to or on the date of cross-over to active treatment with UX003. The change in the number of lines from pre-treatment baseline to 24 weeks of treatment was evaluated. (This provides the valid assessment, as placebo effect would be subtracted from the treatment effect estimate providing a more conservative assessment of the true treatment effect.) A positive change from baseline indicates improvement. Change from baseline in uncorrected visual acuity was analyzed by GEE modeling based on observed data. The GEE model included all participants who had non-missing baseline and at least one post-baseline value during the 24 weeks of UX003 treatment. The model included baseline value, and the UX003 treatment week as a categorical variable. The covariance structure within participants was assumed to be exchangeable.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: lines
Arm/Group | UX003 4 mg/kg
Number analyzed (Participants) | 7
lines
  Left eye | 1 (0.63)
  Right eye | 0.9 (0.51)
Statistical Analysis 1: Comparison: UX003 4 mg/kg; for the left eye; Test type: Superiority; p = 0.1140, GEE; LS Mean = 1.0, 95% CI 2-sided [-0.2 to 2.2]
Statistical Analysis 2: Comparison: UX003 4 mg/kg; for the right eye; Test type: Superiority; p = 0.0906, GEE; LS Mean = 0.9, 95% CI 2-sided [-0.1 to 1.8]

8. Secondary Outcome: Change From Baseline in Bruininks-Oseretsky Test of Motor Proficiency (BOT-2) Scores at UX003 Treatment Week 24
Description: BOT-2 was administered to evaluate treatment-related changes in 4 domains assessing both fine and gross motor function: balance (score 0 to 37), fine motor precision (score 0 to 41), manual dexterity (score 0 to 45), and running speed/agility (score 0 to 52). Higher scores indicate more motor proficiency; a positive change from baseline indicates improvement. Baseline was defined as the last assessment prior to or on the date of cross-over to active treatment with UX003. (This provides the valid assessment, as placebo effect would be subtracted from the treatment effect estimate providing a more conservative assessment of the true treatment effect.) Change from baseline in BOT-2 was analyzed by GEE modeling based on observed data. The GEE model included baseline value, and the UX003 treatment week as a categorical variable. The covariance structure within participants was assumed to be exchangeable.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | UX003 4 mg/kg
Number analyzed (Participants) | 11
units on a scale
  Balance: number analyzed (Participants) | 6
  Balance | 0.8 (0.46)
  Fine motor precision | -0.2 (0.23)
  Manual dexterity | 0.2 (0.21)
  Running speed and agility: number analyzed (Participants) | 5
  Running speed and agility | 0.2 (0.12)
Statistical Analysis 1: Comparison: UX003 4 mg/kg; Scale-BALANCE; Test type: Superiority; p = 0.0883, GEE; LS Mean = 0.8, 95% CI 2-sided [-0.1 to 1.7]
Statistical Analysis 2: Comparison: UX003 4 mg/kg; Scale: FINE MOTOR PRECISION; Test type: Superiority; p = 0.3528, GEE; LS Mean = -0.2, 95% CI 2-sided [-0.7 to 0.2]
Statistical Analysis 3: Comparison: UX003 4 mg/kg; Scale-MANUAL DEXTERITY; Test type: Superiority; p = 0.4094, GEE; LS Mean = 0.2, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 4: Comparison: UX003 4 mg/kg; Scale-RUNNING SPEED AND AGILITY; Test type: Superiority; p = 0.1020, GEE; LS Mean = 0.2, 95% CI 2-sided [0.0 to 0.4]

9. Secondary Outcome: Change From Baseline in Pediatric Quality of Life (PedsQL) Multidimensional Fatigue Scale at UX003 Treatment Week 24
Description: The PedsQL 18-item scale is comprised of 3 dimensions: general fatigue (6 items), sleep/rest fatigue (6 items) and cognitive fatigue (6 items). Each item has a 5-point Likert response scale that is reverse scored and transformed to a 0 to 100 scale with higher scores indicating less fatigue. Baseline was defined as the last assessment prior to or on the date of cross-over to active treatment with UX003. (This provides the valid assessment, as placebo effect would be subtracted from the treatment effect estimate providing a more conservative assessment of the true treatment effect.) Change from baseline in PedsQL total fatigue score was analyzed by GEE modeling based on observed data. The GEE model included all participants who had non-missing baseline and ≥1 post-baseline value during the 24 weeks of UX003 treatment. The model included baseline value, and the UX003 treatment week as a categorical variable. The covariance structure within participants was assumed to be exchangeable.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | UX003 4 mg/kg
Number analyzed (Participants) | 12
units on a scale | 3.4 (2.64)
Statistical Analysis 1: Comparison: UX003 4 mg/kg; Test type: Superiority; p = 0.1953, GEE; LS Mean = 3.4, 95% CI 2-sided [-1.8 to 8.6]

10. Secondary Outcome: Percentage of Individual Clinical Response (ICR) Responders at UX003 Treatment Week 24
Description: Percentage of participants who were ICR responders based on MID criteria at Week 24. At the Randomization visit, the physician queried the participant or parent/caregiver about signs and symptoms of MPS VII that interfered most with the participant's daily life. Answers were mapped to an appropriate clinical outcome measure (e.g., difficulty walking could map to the 6MWT; breathing problems to FVC). The clinical outcome ranked with the highest impact on daily life that could be reliably completed by the participant and met a threshold level of impairment was selected as the ICR for that participant. ICR response was assessed based on a positive change (according to pre-specified MID criteria) of each participant's ICR. Agresti-Coull confidence interval with nominal coverage ≥ 95%.
Time Frame: as for outcome 2
Population: Participants who had non-missing baseline and ≥1 post-baseline value during 24 weeks of UX003 treatment. Given a randomized blind start and single crossover study design, all 4 groups received a minimum of 24 weeks of UX003 treatment, with a placebo period ranging from 0-24 weeks, by group. Analysis of placebo data was not planned.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UX003 4 mg/kg
Number analyzed (Participants) | 12
percentage of participants | 25 [8.3 to 53.8]

11. Secondary Outcome: Change From Baseline in Impactful Clinical Problem Total Score at UX003 Treatment Week 24
Description: The 3 most impactful clinical problems as reported by the subject/parent/caregiver during the Clinical Problem Evaluation were scored on a Likert scale from 1 (very little problem) to 7 (an extreme amount) at randomization and post-randomization visits. At post-randomization visits, each clinical problem was again scored for impact on daily activities. Total scores ranged from 3 to 21; lower scores reflect less impact on daily life. Baseline was defined as the last assessment prior to or on the date of cross-over to active treatment with UX003. (This provides the valid assessment, as placebo effect would be subtracted from the treatment effect estimate providing a more conservative assessment of the true treatment effect.) The change from baseline up to UX003 Treatment Week 24 were analyzed by GEE modeling, including baseline value, and the post-UX003 initiation treatment week as a categorical variable. The covariance structure within participants is assumed to be exchangeable.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | UX003 4 mg/kg
Number analyzed (Participants) | 12
units on a scale | -1.2 (0.92)
Statistical Analysis 1: Comparison: UX003 4 mg/kg; Test type: Superiority; p = 0.2022, GEE; LS Mean = -1.2, 95% CI 2-sided [-3.0 to 0.6]

ADVERSE EVENTS:
Time Frame: Safety information was collected for all participants who received any study drug from signing the informed consent form through 30 days after last dose of study drug. Mean treatment duration for UX003 was 36.0 weeks, and for placebo was 15.8 weeks.
Description: Treatment-emergent adverse events (TEAEs) are presented. Given that the study has only has 12 participants, and a by arm/group analysis would include no more than 3 participants per arm/group, the TEAE summary was planned to present data by treatment only.
Groups:
- Placebo: Participants received placebo for the first 8 weeks (Group B), 16 weeks (Group C) or 24 weeks (Group D) of the study, based on the blind-start design.
- UX003 Active Treatment: Participants received 4 mg/kg UX003 QOW per group assignment (based on the blind-start design) and were dosed through Week 46. All groups received a minimum of 24 weeks of treatment with UX003.
Arm/Group | Placebo | UX003 Active Treatment
Serious Adverse Events (participants affected / at risk) | 0/9 | 2/12
Other Adverse Events (participants affected / at risk) | 9/9 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | UX003 Active Treatment (N=12)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 — CTCAE grade 2 non-related craniocerebral injury as a result of falling off the bed. Computed tomography scan of the head did not show intracranial bleeding nor acute intracranial injury.
Anaphylactoid reaction (Immune system disorders) | 0 | 1 — CTCAE grade 3 treatment-related anaphylactoid reaction secondary to an infusion rate error occurring during the first hour of UX003 administration.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | UX003 Active Treatment (N=12)
Hypertension (Vascular disorders) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaphylactoid reaction (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 1
Infusion site extravasation (General disorders) | 1 | 4
Oedema (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Catheter site bruise (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Infusion site bruising (General disorders) | 0 | 1
Infusion site swelling (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Infusion site discomfort (General disorders) | 1 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Body temperature increased (Investigations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Clonus (Nervous system disorders) | 0 | 1
Dysstasia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abnormal faeces (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Cheilosis (Gastrointestinal disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 5
Ear infection (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days